CLINICAL TRIAL: NCT04000893
Title: Effect of Aerobic or Resistance Exercise on the Endothelial Response in Post-acute Myocardial Infarction Patients Submitted to Angioplasty: Randomized Clinical Trial
Brief Title: Effect of Aerobic or Resistance Exercise on the Endothelial Response in Post-acute Myocardial Infarction Patients Submitted to Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AMI and exercise
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Cardiac Rehabilitation; Aerobic Exercise; Resistance Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise session (Experimental): Acute isometric session, about 20 minutes.
  Interventions: Other: Resistance exercise session
- Aerobic exercise session (Active Comparator): Acute aerobic session, about 20 minutes.
  Interventions: Other: Resistance exercise session

INTERVENTIONS:
Other: Resistance exercise session — Acute isometric exercise session performed with handgrip Jamar about 20 minutes monitored.
  Other Names: Aerobic exercise session

SUMMARY:
Cardiac Rehabilitation, as art and acting science multiprofessional, is based on the training with exercises that provides the post-infarct patients to satisfactorily re-establish the patient's clinical condition and that improve the functional capacity of these individuals.

Evidence shows that aerobic exercise training provides improvements in the endothelial function of this population. However, we do not yet have strong evidence of other modalities of exercise in these parameters in post-infarction patients treated with angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Post-acute myocardial infarction patients
* Ergometric test 30 days after the infarction
* Ejection fraction> 40% (Simpson's method)
* Regular use of optimized drugs

Exclusion Criteria:

* Unable to perform the randomized exercise

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Pre and post 5 minutes exercise session
  Flow-mediated dilatation technique

SECONDARY OUTCOMES:
Arterial stiffness | Pre and post 5 minutes exercise session
  Pulse wave velocity technique

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lehnen, PhD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Alexandre Lehnen, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kollet DP, Marenco AB, Belle NL, Barbosa E, Boll L, Eibel B, Waclawovsky G, Lehnen AM. Aerobic exercise, but not isometric handgrip exercise, improves endothelial function and arterial stiffness in patients with myocardial infarction undergoing coronary intervention: a randomized pilot study. BMC Cardiovasc Disord. 2021 Feb 17;21(1):101. doi: 10.1186/s12872-021-01849-2. PMID 33596832